CLINICAL TRIAL: NCT07016503
Title: Investigation of the Effect of Professional Values Education on Pediatric Nurses' Perception of Professional Values, Emotional Labor Behavior and Burnout Level: A Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of Professional Values Education in Pediatric Nurses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Nazmiye Yirik, graduate student, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14/204
Record Dates: First submitted 2025-05-25; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Nurse Training; Nurse; Professional Burnout; Professional Values
Keywords: Professional values; Professional burnout; Emotional labor; Pediatric nurse; Training program
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): A half-day training plan consisting of three sessions was applied face to face to the nurses in this group at the conference hall of the hospital where the study was conducted on a date determined jointly by the participants and the hospital management (Table 1). Before the training, the nurses in the intervention group were divided into two groups (first group: 17, second group: 18 people) and half-day training was given to one group in the morning and the other group in the afternoon. Since our research is a study evaluating the effectiveness of the training, all training content was provided for the use of the nurses in the intervention group via the website for three months.In order to achieve this, the participating nurses were able to access the training materials with the username and password given to them. During this three-month period, reminder messages such as using the website content, sending update notifications, and sharing spot information and videos regarding profess
  Interventions: Other: Professional values education
- Control group (No Intervention): No intervention was applied to the participants in this group within the scope of the research. After the post-test application of the research, this group was also given the same training as the intervention group, independent of the research, and the website was opened for use.

INTERVENTIONS:
Other: Professional values education — At this stage, a comprehensive literature review was conducted and professional values education was prepared. The prepared education content was transferred to a website for which a domain was purchased within the scope of the research. The developed website was presented to the opinion of a group of 7 experts in terms of content: Child Health and Diseases Nursing Department Faculty Members (4), Nursing Fundamentals Department Faculty Members (1), Public Health Nursing Department Faculty Members (2). Expert opinions were evaluated with the measurement tool prepared by the researchers in line with the literature.
  Arms: experimental group

SUMMARY:
H1. 1: The professional values perception level of pediatric nurses who received professional values education significantly increases compared to the control group.

H1. 2: The surface behavior score of emotional labor strategies of pediatric nurses who received professional values education significantly decreases compared to the control group.

H1. 3: The deep behavior score of emotional labor strategies of pediatric nurses who received professional values education significantly increases compared to the control group.

H1. 4: The sincere behavior score of emotional labor strategies of pediatric nurses who received professional values education significantly increases compared to the control group.

H1. 5: The burnout/emotional exhaustion levels of pediatric nurses who received professional values education significantly decreases compared to the control group.

H1. 6: The desensitization/cynicism levels of pediatric nurses who received professional values education significantly decreases compared to the control group.

H1. 7: The personal success levels of pediatric nurses who received professional values education significantly increase compared to the control group.

DETAILED DESCRIPTION:
In recent years, the rapid advancement of technology in the field of health has led to changes in the needs and expectations of society, and the importance of professional values in the nursing profession, which has an important role for society, has been increasing (Lee et al., 2020; Bijani et al., 2019). Nursing is a discipline that has undergone various changes from past to present, with the main goal of protecting and improving the health of individuals, families and society. The nursing profession, which initially focused only on physical health, has expanded its perspective over the years and has adopted a holistic approach to individuals in terms of physical, spiritual and sociocultural aspects (Göriş et al., 2014). In addition to these, professional responsibilities have increased (Bijani et al., 2019), it has become autonomous and has aimed to improve health as well as prevent diseases (Göriş et al., 2014). Experience has begun to give way to professionalism in nursing (Tüfekçi, 2015). Professional nurses are nurses who follow scientific developments, have high autonomy, and embrace professional and ethical values. In this respect, nurses constitute the evolving role of the profession. Professional values are the basic principles and beliefs that guide professional groups in their own fields of decision-making and practice (Weis & Schank, 2002). In addition, it is stated that professional values form the basis of nursing practice (Poorchangizi et al., 2019). In the field of pediatric nursing, where different age groups are included, care needs vary to the same extent. Pediatric nurses are responsible for effectively coping with the reactions of children to illness, developmental crises during the illness, and problems caused by the illness according to age groups (Shuck et al., 2013). The acquisition of professional values in this field and their transfer to practice is an important component that contributes to the development of the profession. Children cared for by pediatric nurses cannot make their own decisions. In situations where decisions need to be made, the family must make the decision. This situation sometimes causes ethical dilemmas (Griffin et al., 2021). It should not be forgotten that nurses can solve these ethical dilemmas by resorting to professional values (Poorchangizi et al., 2019). Pediatric nurses provide quality care to their patients with the professional values they have (Poreddi et al., 2021). Nurses who spend the most time with patients and provide primary care experience various emotions due to the nature of their profession. During this care and application process, nurses are expected to show emotions such as empathy, compassion, and interest, while they are expected to avoid negative emotions such as anger and disappointment (Hwang & Park, 2022). It is stated that nurses' emotions are an important element in their relationships with their patients, and it is emphasized that they will be effective in the recovery process of patients (Lee & Jang, 2019).In addition to professionalism, pediatric nurses carry a great emotional burden due to their responsibilities such as caring for children with chronic diseases, experiencing ethical dilemmas, and supporting the child and their family (Griffin et al., 2021). Nurses demonstrate emotional labor behavior in order to understand and successfully manage emotions such as pain, suffering, fear, and anxiety felt by children (Öz & Baykal, 2017; Aydın et al., 2019). Emotional labor is defined as exhibiting an appropriate stance for the situation, regardless of the actual emotion. In other words, it is the energy spent by employees to hide emotions that are inappropriate for the situation and display emotions that are appropriate (Humphrey, 2021; Masracci & Adams, 2019). Studies have shown that emotional labor negatively affects the health of employees. Musculoskeletal problems, burnout, and depression are the main ones (Ha et al., 2021; Guajardo & Vasquez, 2018). In addition, pediatric nurses receive comprehensive medical training throughout their education, but they often lack emotional and psychological training.This situation leads to burnout in pediatric nurses (Restrepo & Pilgrim, 2011; Altan & Özpehlivan, 2019). Pediatric nurses are pioneers in providing non-traumatic, compassionate care with a family-centered care philosophy. Studies have recommended the development of training programs to strengthen professional values and emotional labor behavior in pediatric nurses (Freitas et al., 2021; Youn and Nouh, 2018). In addition, it is stated that professional values positively affect areas such as job satisfaction (Kootahi et al., 2023; Kaya, 2019), family involvement in care (Demirci, 2019), caring behaviors (Güven, 2021; Bekleviç, 2019; Bulut & Kızılırmak, 2022; Şanal, 2020), and patient safety (İşeri & Sarıtaş, 2023). All these concepts constitute the components of professional values. In this context, the purpose of our research is to examine the effect of professional values education on pediatric nurses' perception of professional values, emotional labor behavior and burnout level.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in a pediatric clinic Nurses who volunteer

Exclusion Criteria:

* Nurses working outside of the pediatric clinic Non-volunteer nurses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Nurses' professional values scale nurses' emotional labor behavior scale Maslach burnout scale | January 2024-January 2025
  Nurses' professional values scale nurses' emotional labor behavior scale Maslach burnout scale

CONTACTS AND LOCATIONS:
Locations (1):
- Isparta City Hospital, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yirik N, Tutar S. Investigation of professional values education's effect on pediatric nurses' perception of professional values, emotional labour behaviours and burnout levels: A randomised controlled trial. J Pediatr Nurs. 2026 Jan 9;87:99-110. doi: 10.1016/j.pedn.2025.12.030. Online ahead of print. PMID 41518791
- See also: Related Info — http://www.hemsireliktedegerler.com